CLINICAL TRIAL: NCT02198157
Title: Effect of Intermittent Versus Continuous Bladder Catheterization During Labor on Second Stage Duration
Brief Title: Urinary Catheterization and Second Stage of Labor
Acronym: cath2stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raed Salim (Other)
Responsible Party: Sponsor-Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45-14-EMC
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Labor, Second Stage
Keywords: duration of second stage; urinary catheterization; epidural anaesthesia
MeSH Terms: interventions — Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intermittent urinary catheterization (Active Comparator): nullipara women with epidural anaesthesia who pose urination difficulty will receive intermittent catheterization
  Interventions: Other: urinary catheterization
- continuous urinary catheter (Active Comparator): nullipara women with epidural anaesthesia who pose urination difficulty will receive continuous catheterization
  Interventions: Other: urinary catheterization

INTERVENTIONS:
Other: urinary catheterization — nullipara women with epidural anaesthesia who pose urination difficulty will be randomize to receive intermittent or continuous urinary catheterization.
  Other Names: continuous versus intermittent catheterization.

SUMMARY:
* Labor is divided into three stages: the first stage is from labor onset until full dilation, second stage is from full dilation until delivery of the baby, and the third stage from the delivery of the baby until the delivery of the placenta
* The mean duration of second stage in nulliparas as defined by the American college of obstetricians and gynecologists (ACOG) is 54 minutes
* Epidural anesthesia is a known cause for prolongation of the second stage of labor. Prolonged second stage in nullipara women with epidural is defined as more than 3 hours, and more than 2 hours in those without epidural.
* Although perinatal outcome is not compromised with a prolonged second stage , there is evidence that maternal morbidities such as perineal trauma, chorioamnionitis ,instrumental delivery and postpartum hemorrhage increase with prolonged second stage
* Another effect of epidural anesthesia during labor is urinary retention and a need for catheterization.
* Full bladder may behave as a tumor previa and interfere to fetal head descent in the birth canal, increasing by that the duration of the second stage.
* This study aims to investigate the effect of intermittent versus continuous catheterization on the duration of the second stage of labor

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Gestational age 24-42 weeks
* epidural anaesthesia
* Vertex presentation
* Singleton

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
duration of second stage of labor | within the first 48 hours after delivery

SECONDARY OUTCOMES:
chorioamnionitis | within the first 48 hours after delivery

OTHER OUTCOMES:
post-partum hemorrhage | within the first 48 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: raed salim, MD, Study Director — Dep. OB/GYN, HaEmek Medical Center, Afula, Israel; abeer suleiman, MD, Principal Investigator — Dep. OB/GYN, HaEmek Medical Center, Afula, Israel
Locations (1):
- Dep. OB/GYN, HaEmek Medical Center, Afula, Israel